CLINICAL TRIAL: NCT03350594
Title: Family Therapy and Anorexia Nervosa : Which is the Best Approach? Family Therapy Multicenter Randomised Control Trial of Systemic Family Therapy Versus Multiple Family Therapy
Brief Title: Family Therapy and Anorexia Nervosa : Which is the Best Approach?
Acronym: THERAFAMBEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Mutualiste Montsouris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); PHRC Interrégionnal 2015 (Unknown); Fondation Sandrine Castellotti (Unknown); Fondation de l'Avenir (Other); CESP - UMR 1018 / INSERM (Unknown); Direction Générale de l'offre de Soins (DGOS) (Unknown); University Hospital, Rouen (Other); Maison des Adolescents de Cochin (APHP) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY-2016-01; 2016-A00818-43 (Other: IDRCB Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa; Multiple Family Therapy; Systemic Family Therapy; Adolescence; Randomised controled trial
MeSH Terms: conditions — Anorexia Nervosa | interventions — Psychotherapy, Group

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic Family Therapy (Active Comparator): SyFT involves the patient, the parents, and siblings over the age of 6 living at home. Therapists do not manage the issues relating to AN, which are taken on by referent psychiatrist who can be called on in case of any concern. Without denying personal suffering and its intra-psychic and meta-psychological impact, or the somatic and biological aspect of the pathology, the emphasis is on interactions around the symptom.
  There will be free exchanges along the lines between therapist and family, within the family and between therapists.
  Session is possible with sibling alone or the parents alone or in inter-generational mode (other family relatives)
  Interventions: Behavioral: Systemic Family Therapy
- Multiple Family Therapy (Experimental): Each session will involve 5 families of patients suffering from AN including the parents and non-systematically the siblings. There will be exchanges in groups and mediation via different exercises involving different sub-groups according to the theme: complete families, patients on their own for problems specific to them, or " cross-parenting " exercises whereby parents adopt another patient for the duration of the exercise. This organization enables mutual support and social propping, favoring the emergence of family resources. Direct exchanges between families (between parents, siblings, or mixes) with and between therapists are also sought.
  Interventions: Behavioral: Multiple Family Therapy

INTERVENTIONS:
Behavioral: Systemic Family Therapy — Patient will have 10 sessions of Systemic Family Therapy during 12 months with his/her family.
  Arms: Systemic Family Therapy
Behavioral: Multiple Family Therapy — Patient and his/fer family will have 10 sessions of Multiple Family Therapy during 12 months.
  Arms: Multiple Family Therapy

SUMMARY:
The aim of this study is to evaluate whether the implementation of Multiple Family Therapy (MFT) within a multi-disciplinary treatment program for Anorexia Nervosa (AN) in adolescence is at least as effective in terms of clinical Body Mass Index evolution as single Systemic Family Therapy (SyFT) after 12 months of treatment. We expect that these two techniques will not differ in terms of global efficacy, but that MFT could be more suitable for certain profiles who may be less responsive to SyFT.

DETAILED DESCRIPTION:
While family therapy is considered to have proved itself, its efficacy has been tested with reference to individual therapy by several teams of researchers or in addition to an overall treatment program. Few studies however have compared different types of family studies, and these studies were often on small samples. In addition, efficacy in terms of remission at 12-18 months was below 50% for large samples, and whatever the technique envisaged. Consequently, there is a need for exploration of this type of care provision. It is in this context, and also on account of budget considerations, to avoid hospitalizations, that the Maudsley team developed MFT for AN in the form of intensive day-care. The system is open to debate (there is a selection of highly motivated subjects able to suspend family and professional activities for some 20 days a year, and to find accommodation close to the hospital, and ready to relinquish other types of follow-up. However, MFT is, according to its advocates (families, caregivers) a therapeutic tool that is effective and appreciated by families. Other teams have therefore adapted it to care practices in France, and suited it to children, adolescents or adult in ambulatory care. In addition, we are aware that our care program is not satisfactory (fewer than half the subjects are cured after 12 to 18 months of treatment) and hence perfectible. We would like to use MFT, but this approach, particularly in ambulatory setting, has never been evaluated in comparison with another type of therapy in a randomized trial. We therefore wish to perform a randomized controlled trial to assess the contribution of MFT to the treatment of AN in comparison with SyFT.

The project is original in that, for the first time, it sets out to assess MFT in adolescent AN in ambulatory care in reference to SyFT, to estimate cost parameters relating to the two techniques, and also to identify the profiles of the best responders according to patient characteristics.

Family therapy will be established either after first half of hospitalization (half way to weight gain fixed for discharge), or when the patient seen in consultation is in a stable clinical state with no indication for hospitalization.

Patient will be randomized to MFT or SyFT after agreement to take part in the study. Randomization will be stratified on care provision status at inclusion (ambulatory or hospitalized - the latter being a possible selection bias according to severity) and therapies will start in the month following the randomization.

Patients and their families will have one session a month MFT ou SyFT during 12 months.

Evaluations will take place at the end of therapy at 12 months, then at the 6 months follow-up. Evaluators will be blind to the treatment group and will use a standardized research questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from Anorexia Nervosa according to DSM-5 criteria (restricting or purge type Anorexia Nervosa)
* Patient with the paucisymptomatic form of Anorexia Nervosa
* Patient suffering from Anorexia Nervosa before his 19 years old
* Patient aged between 13 and 19
* Patient and his/her parents who accept to participate to the study
* Patient and his/her parents who live in Paris or Rouen and surroundings

Exclusion Criteria:

* Patient who is diagnosed with: psychosis, mentale deficiency, organic cerebral disorder, any pathology that interfere with feeding or its regurgitation
* Patient who does not speak french
* Patient who is already followed in a familial therapy

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2023-11-11 (Estimated); Study Completion 2024-05-10 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | Baseline, 12 months
  Change from baseline Body Mass Index (Weight in KG / Height in m²) at 12 months

SECONDARY OUTCOMES:
Change from Baseline overall clinical outcome at 12 months and 18 months | Baseline, 12 months, 18 months
  Assess with the Morgan and Russell outcome categories. A quantitative score (0-12) was obtained through four subscales: Food intake, Menstrual state, Mental state, Psychosexual state and Socioeconomic state. The higher the score, the better the clinical state.
  We use BMI percentiles that are a good relevant index. Hence, to take the ages of our patients into account, we refer to the INSERM (French National Institute for Health and Medical Research) weight curves for the French population, in which a BMI 10th percentile indexes AN.
  We define the Morgan and Russell outcome categories as follows: 1) Good outcome: weight>10th BMI percentile and regular menstruation; 2) Intermediate outcome: weight>10th BMI percentile but amenorrhea (i.e., the absence of menstruation for at least the past three months); 3) Poor outcome: weight <10th BMI percentile and/or presence of bulimic symptoms.
  We will pool the Good and Intermediate outcome categories.
Change from baseline nature and seriousness of eating-disorder symptoms at 12 months and 18 months | Baseline, 12 months, 18 months
  Patients will complete the Eating Disorder Inventory-2 (EDI-2) and the Eating Disorder Diagnostic Scale (EDDS) to assess their current eating disorder (ED) symptomatology. The EDI-2 consists of 91 questions that make up 11 subscales measuring ED pathology and psychopathology. A higher total score represents a higher burden of disease level of symptomatology. The EDDS is a 22-item questionnaire measuring anorexia nervosa, bulimia nervosa and binge eating disorder. The scale consists of a combination of Likert scores (ranging from 0 (not at all) to 6 (extremely)), dichotomous scores, frequency scores and open-ended questions like weight and height. It is a diagnostic scale and a symptom composite scale. An overall eating disorder symptom composite score is computed by standardizing and summing up scores across all items.
Change from baseline patient's Emotional symptoms at 12 months and 18 months | Baseline, 12 months, 18 months
  Several criterias will be evaluate to assess patient's emotional symptoms, using the following questionnaires : HADS (Hospital Anxiety and Depression Scale) and BID-13 (Beck Depressive Inventory-13) to evaluate anxiety and depression, BVAQ-B (Bermond-Vorst Alexithymia Questionnaire) to evaluate alexithymic features, MOCI (Maudsley Obsessional-Compulsive Inventory) to evaluate obsessive-compulsive symptoms, LSAS-CA (Liebowitz Social Anxiety Scale for Children and Adolescents) to measure social anxiety, RES (Rosenberg Self-Esteem) to measure self-esteem, OSI (Ottawa Self-Injury) to measure occurrence, frequency, level of motivation to stop, types and functions and potential addictive features of self-injury, and C-SSRS (Columbia-Suicide Severity Rating Scale) to distinguish the domains of suicidal ideation and suicidal behaviour.
Change from baseline parent's Emotional symptoms at 12 months and at 18 months | Baseline, 12 months, 18 months
  Several criterias will be evaluate to assess parent's emotional symptoms using the following questionnaires : HADS (Hospital Anxiety and Depression Scale) and BID-13 (Beck Depressive Inventory-13) to evaluate anxiety and depression, BVAQ-B (Bermond-Vorst Alexithymia Questionnaire) to evaluate alexithymic features, RES (Rosenberg Self-Esteem) to measure self-esteem, ECI (Experience Caregiving Inventory) to measure the experience of caring for an individual with a severe mental illness, EDSIS (Eating Disorders Symptom Impact Scale) to measure caregiving burden in eating disorder, MIV-TIG (Mental Illness Version of Texas Inventory Grief) to measure past and current feeling of loss in relatives of people suffering of mental illness.
Change from baseline quality of family relationships at 12 months and 18 months | Baseline, 12 months, 18 months
  The following questionnaires will be used to assess the family relationships : the Score-15, a self-report outcome measure designed to be sensitive to the kinds of changes in family relationships, and the FAD (Family Assessment Advice) to measure structural, organizational, and transactional characteristics of families.
  Patient will also complete the LEE (Level of Expressed Emotion) while the parents will complete the FQ (Family Questionnaire) assessing the expressed emotion status (criticism, emotional, over-involvement) of relatives of patients.
Change from baseline patient's quality of life at 12 months and at 18 months | Baseline, 12 months, 18 months
  We will use the Eating Disorders Quality of Life Questionnaire (EDQOL) and the Social and Occupational Functioning Scale (SOFAS) for patients.
  The EDQOL has 25 items that contribute to four subscales (Psychological, Physical/Cognitive, Work/School, and Financial), which combined produce an overall quality of life score. Each item is coded on a five-point scale and asks the participant to rate the extent to which they perceive their eating disorder to affect their quality of life in different domains. Higher scores indicate lower quality of life.
  The SOFAS is a rating scale used to subjectively assess the social and occupational functioning due to medical conditions. The scale is based on a continuum of functioning, ranging from 0 to 100, with higher scores indicating better functioning.
Change from baseline parent's quality of life at 12 months and at 18 months | Baseline, 12 months, 18 months
  Parents will answer the following questionnaires:
  The WHOQOL (World Health Organization Quality of Life) to evaluate quality of life that can be defined as an individual's subjective perception of different aspects of life that are influenced by health status and includes subjective evaluations of physical functioning, mental health, and social/role functioning.
  The LHS (the London Handicap Scale) to determine the effect of chronic disorders on a person's functional ability using a self-completion questionnaire. Each degree of handicap along a 6-point interval was assigned a scale weight. Six scales are rated Mobility, Physical independence : Occupation ; Social integration: Orientation, Economic self-sufficiency. A total score from 0 to 1 and lower score indicate total disability.
  The CarerQoL-7D (Care-related Quality of life) to describe caregiver burden in seven dimensions (ie, fulfillment, relational, mental, social, financial, perceived support, and physical).
Change from 12-month Patient and parent satisfaction at 18 months | 12 months, 18 months
  Patients and parents will complete quantitative measures: a modified version of the CSQ-8 (Client Satisfaction Questionnaire-8) and a purpose-designed satisfaction interview assessing client satisfaction with a service.

OTHER OUTCOMES:
Change from baseline Cost-efficiency analysis at 12 months and 18 months | 12 months, 18 months
  Total cost of treatment calculated by aggregating the health care consumption recorder by the french health insurance system

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin CARROT, MD, Principal Investigator — Institut Mutualiste Montsouris
Locations (5):
- France (5):
  - Hôpital Salvator - APHM Marseille, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Institut Mutualiste Montsouris, Paris
  - Maison de Solenn - Maison des Adolescents Cochin, Paris
  - Clinique Médicale et Pédagogique Edouard RIST, Paris

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carrot B, Duclos J, Barry C, Radon L, Maria AS, Kaganski I, Jeremic Z, Barton-Clegg V, Corcos M, Lasfar M, Gerardin P, Harf A, Moro MR, Blanchet C, Godart N. Multicenter randomized controlled trial on the comparison of multi-family therapy (MFT) and systemic single-family therapy (SFT) in young patients with anorexia nervosa: study protocol of the THERAFAMBEST study. Trials. 2019 Apr 30;20(1):249. doi: 10.1186/s13063-019-3347-y. PMID 31039797